CLINICAL TRIAL: NCT04043364
Title: LIVE@Home.Path: a Mixed Method, Stepped Wedge and Randomized Controlled Trial Innovating the Clinical Pathway for Home-dwelling Persons With Dementia and Their Families
Brief Title: Live@Home.Path: Innovating the Clinical Pathway for Home Dwelling Persons With Dementia and Their Families
Acronym: LIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Bergen (Other)
Collaborators: Haraldsplass Deaconal Hospital (Unknown); Western Norway University of Applied Sciences (Other); Norwegian Reseach Centre AS (NORCE) (Unknown); Norwegian National Advisory Unit on Ageing and Health (Unknown); Natioal Association for Public Health (Unknown); Municipality of Bergen (Unknown); Municipally of Kristiansund (Unknown); Municipally of Bærum (Unknown); The Dignity Centre (Unknown); Harvard McLean University (Unknown); Yale University (Other); University College, London (Other); University of Leiden (Unknown); Tohoku University (Other); King's College London (Other); The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: NFR 273581
Record Dates: First submitted 2019-03-15; First posted 2019-08-02 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-01

CONDITIONS: Dementia; Home-dwelling; Caregiver
Keywords: Learning; Innovation; Volunteers; Empowerment
MeSH Terms: conditions — Dementia; Empowerment

STUDY DESIGN:
Intervention Model Description: Mixed method, stepped wedge randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIVE (Experimental): A multicomponent intervention focusing on Learning, Innovation, Volunteers and Empowerment organized by a local coordinator.
  Interventions: Behavioral: LIVE
- Treatment as usual (No Intervention): Care coordination and facilitation as usual.

INTERVENTIONS:
Behavioral: LIVE — Learning, Innovation, Volunteers and Empowerment
  Arms: LIVE

SUMMARY:
This study aims at developing, implementing and evaluating a complex intervention involving Learning, Innovation, Volunteers and Empowerment for home dwelling persons with dementia and their caregivers. The investigators hypothesise that a successfully implemented intervention will reduce caregivers burden and be cost-effective.

DETAILED DESCRIPTION:
The provision of economically viable and proper care for the growing group of home-dwelling people with dementia (PWD) is one of the most pressing issues in our society. While a cure for dementia is not yet available, professionals and policy-makers highly prioritize the support of caregivers who experience a vast burden. However, there is a lack of high-quality research investigating clinical, social and economic factors that may add beneficial effects. This project aims to develop, test, and implement a complex intervention for PWD, intended to reduce caregivers' burden, which will aid PWD to stay safely, longer and independently at home with dignity and cost-effectiveness. The term informal caregivers' burden may include different meanings for different people and be related to economic burden, depression and anxiety, quality of life (QoL), or simply the quality of sleep and recreation. In a stepped wedge, cluster randomized controlled trial, involving primary and secondary health care systems in Bergen, Bærum and Kristiansand the 24-month LIVE@Home.Path study will be undertaken in a stepped wedge design. The user-inspired and tailored intervention includes a designated coordinator to the PWD and caregiver for 6 months to introduce a complex intervention involving a) Learning b) Innovation c) Volunteers and d) Empowerment.

Qualitative interviews will determine users' values and wishes, and promotors and barriers for successful implementation of the intervention. Primary and secondary outcomes on cognitive, emotional and social factors, cost-benefit analyses, and QoL of PWD and families will be assessed every 6-month over 2 years.

Update spring 2020: The COVID-19 pandemic severely hampered the implementation of the intervention for the second group. We therefore had to change the design, postponing the intervention in Bærum and Kristiansand, and delivering the intervention in Bergen by phone. In addition, we initiated the PAN.DEM in the LIVE@Home.Path trial, collecting data from phone interviews with caregivers on change in Health services and neuropsychiatric symptoms, risk perception and restrictions. Changes in design approved by Ethical committee (REK: 10861).

ELIGIBILITY:
Inclusion Criteria:

1. Home-dwelling people with dementia (PWD) equal or above 65 years diagnosed according to national guidelines
2. Mini mental state examination score 15-24
3. Functional Assessment Staging Test (FAST score 4-7)
4. Living with a partner, or have regular contact with a caregiver minimum 1 hour/week

Exclusion Criteria:

1. Participate in other trials
2. Expected survival under 4 weeks

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 280 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Resource Utilization in Dementia | up to 24 months follow up, assesment every 6 months
  RUD:A validated tool for assessment of time use for cost effectiveness analyses, measuring total time use in hours/day for different activities, numbers of contact points with care professionals and use of medications, high time use, many contacts and many medications indicates high resource use
Relative stress scale | up to 24 months follow up, assessment every 6 months
  RSS: measuring caregiver distress, 15 items ranging from 0-4, high score indicates high burden

SECONDARY OUTCOMES:
Activities of daily living, instrumental | 24 months follow up, assesment every 6 months
  I-ADL scale assessing instrumental activities such as use of telephone, economy, household, public transport and shopping, range from 8-31, higher score indicates poorer functioning
Depression and mood | 24 months follow up, assesment every 6 months
  CSDD: Cornell scale for depression in dementia, range 0-38, high score indicates high symptom load
Agitation | 24 months follow up, assesment every 6 months
  CMAI: Cohen-Mansfield Agitation Inventory, 29 items assessing the frequency of agitated behaviour, range 29-203, high score indicates higher severity
Neuropsychiatric symptoms | 24 months follow up, assesment every 6 months
  NPI: presence, severity and burden of depression, anxiety, psychosis and motor disturbances, range from 0-144, high score indicates frequent, severe and burdensome symptoms
Adverse events | 24 months follow up, assesment every 6 months
  Falls, disappearances outdoor, admissions to acute wards, fire hazard
Use of assistive technology | 24 months follow up, assesment every 6 months
  number of technical aids, cognitive intervention devices and assisted-living systems
Use of volunteers | 24 months follow up, assesment every 6 months
  number of participants with contact with a volunteer, number of hours spent with volunteer
Activities of daily living, personal | 24 months follow up, assesment every 6 months
  P-ADL, assessing personal activities such as toileting, grooming, dressing, transfer and eating, scale range 6-30, higher score indicates poorer personal functioning
Quality of Life | 24 months follow up, assesment every 6 months
  EQ-5D-5L, Descriptive measure of health related quality of life comprising 5 Dimensions With 5 Levels each, scores can be converted to a single summary index number
Quality of Life VAS scale | 24 months follow up, assesment every 6 months
  EQ-5D, Descriptive measure of quality of life rated on a VAS scale range 0-100, high score indicates good health
Quality of Life | 24 months follow up, assesment every 6 months
  QoL-AD: Quality of life in Alzheimer dementia, 13 items likert scale, range from 13-52 points, high score indicates high quality of life
Use of volunteers | 24 months follow up, assesment every 6 months
  number of hours spent with a volunteer
Change achieving | at the start of intervention, and every 6 months
  Clinical global impression of change, to quantify and track patient progress and treatment response on a scale from 1 to 7, at which 7 indicates substantial worsening.
Caregiver depression | 24 months follow up, assesment every 6 months
  GDS: Geriatric depression scale, 30 items rated yeas or no, high score indicates high burden
Comorbidity | 24 months follow up, assesment every 6 months
  GMHR: General medical health rating scale, 4 point likert scale, range from 1-4, high score indicates high comorbidity burden
Pain in dementia | 24 months follow up, assesment every 6 months
  MOBID-2: assesses the intensity of pain based on interpretation of pain related behaviour, range from 0-10, high score indicates high pain intensity
Change in cognitive performance | Baseline
  IQ CODE: Proxy rater instrument for assessment of change in cognitive performance the last 10 years, range 16-80, high score indicates great decline
Medication use | At the start of the intervention, and every 6 onth follow up
  Self and proxy reported use of medications, both regular and on demand
Participation in educational programs | 24 months follow up, assessment every 6 months
  Participation in educational programes, both for persons with dementia and for caregivers.

OTHER OUTCOMES:
COVID-19: risk perception | month 6 to month 12 (during COVID-19 lock down in Norway)
  Caregivers perception of risk of contamination With Sars-Cov-10
COVID-19: restrictions | month 6 to month 12 (during COVID-19 lock down in Norway)
  Change in services and contact due to restrictions of COVID-19
COVID-19: caregiver burden | month 6 to month 12 (during COVID-19 lock down in Norway)
  Caregivers perception of caregiver burden during COVID-19
COVID-19: neuropsychiatric symptoms | month 6 to month 12 (during COVID-19 lock down in Norway)
  NPI: change in presence, severity and burden of depression, anxiety, psychosis and motor disturbances
COVID-19: depression and mood | month 6 to month 12 (during COVID-19 lock down in Norway)
  CSDD: Change in cornell scale for depression in dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Husebø, MD, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
We plan to make individual participant data available to collaborators and researchers affiliated with the project.

REFERENCES:
- [Background] Husebo BS, Allore H, Achterberg W, Angeles RC, Ballard C, Bruvik FK, Faeo SE, Gedde MH, Hillestad E, Jacobsen FF, Kirkevold O, Kjerstad E, Kjome RLS, Mannseth J, Naik M, Nouchi R, Puaschitz N, Samdal R, Tranvag O, Tzoulis C, Vahia IV, Vislapuu M, Berge LI. LIVE@Home.Path-innovating the clinical pathway for home-dwelling people with dementia and their caregivers: study protocol for a mixed-method, stepped-wedge, randomized controlled trial. Trials. 2020 Jun 9;21(1):510. doi: 10.1186/s13063-020-04414-y. PMID 32517727
- [Background] Gedde MH, Husebo BS, Erdal A, Puaschitz NG, Vislapuu M, Angeles RC, Berge LI. Access to and interest in assistive technology for home-dwelling people with dementia during the COVID-19 pandemic (PAN.DEM). Int Rev Psychiatry. 2021 Jun;33(4):404-411. doi: 10.1080/09540261.2020.1845620. Epub 2021 Jan 8. PMID 33416012
- [Background] Angeles RC, Berge LI, Gedde MH, Kjerstad E, Vislapuu M, Puaschitz NG, Husebo BS. Which factors increase informal care hours and societal costs among caregivers of people with dementia? A systematic review of Resource Utilization in Dementia (RUD). Health Econ Rev. 2021 Sep 18;11(1):37. doi: 10.1186/s13561-021-00333-z. PMID 34536149
- [Background] Puaschitz NG, Jacobsen FF, Mannseth J, Angeles RC, Berge LI, Gedde MH, Husebo BS. Factors associated with access to assistive technology and telecare in home-dwelling people with dementia: baseline data from the LIVE@Home.Path trial. BMC Med Inform Decis Mak. 2021 Sep 15;21(1):264. doi: 10.1186/s12911-021-01627-2. PMID 34525979
- [Background] Vislapuu M, Angeles RC, Berge LI, Kjerstad E, Gedde MH, Husebo BS. The consequences of COVID-19 lockdown for formal and informal resource utilization among home-dwelling people with dementia: results from the prospective PAN.DEM study. BMC Health Serv Res. 2021 Sep 22;21(1):1003. doi: 10.1186/s12913-021-07041-8. PMID 34551783
- [Background] Husebo BS, Berge LI. Intensive Medicine and Nursing Home Care in Times of SARS CoV-2: A Norwegian Perspective. Am J Geriatr Psychiatry. 2020 Jul;28(7):792-793. doi: 10.1016/j.jagp.2020.04.016. Epub 2020 Apr 22. No abstract available. PMID 32381282
- [Background] Husebo BS, Heintz HL, Berge LI, Owoyemi P, Rahman AT, Vahia IV. Sensing Technology to Monitor Behavioral and Psychological Symptoms and to Assess Treatment Response in People With Dementia. A Systematic Review. Front Pharmacol. 2020 Feb 4;10:1699. doi: 10.3389/fphar.2019.01699. eCollection 2019. PMID 32116687
- [Background] Gedde MH, Husebo BS, Mannseth J, Kjome RLS, Naik M, Berge LI. Less Is More: The Impact of Deprescribing Psychotropic Drugs on Behavioral and Psychological Symptoms and Daily Functioning in Nursing Home Patients. Results From the Cluster-Randomized Controlled COSMOS Trial. Am J Geriatr Psychiatry. 2021 Mar;29(3):304-315. doi: 10.1016/j.jagp.2020.07.004. Epub 2020 Jul 11. PMID 32753339
- [Background] Faeo SE, Bruvik FK, Tranvag O, Husebo BS. Home-dwelling persons with dementia's perception on care support: Qualitative study. Nurs Ethics. 2020 Jun;27(4):991-1002. doi: 10.1177/0969733019893098. Epub 2020 Jan 27. PMID 31986964
- [Background] Faeo SE, Tranvag O, Samdal R, Husebo BS, Bruvik FK. The compound role of a coordinator for home-dwelling persons with dementia and their informal caregivers: qualitative study. BMC Health Serv Res. 2020 Nov 16;20(1):1045. doi: 10.1186/s12913-020-05913-z. PMID 33198779
- [Background] Faeo SE, Husebo BS, Bruvik FK, Tranvag O. "We live as good a life as we can, in the situation we're in" - the significance of the home as perceived by persons with dementia. BMC Geriatr. 2019 Jun 6;19(1):158. doi: 10.1186/s12877-019-1171-6. PMID 31170916
- [Background] Gedde MH, Husebo BS, Mannseth J, Naik M, Selbaek G, Vislapuu M, Berge LI. The impact of medication reviews by general practitioners on psychotropic drug use and behavioral and psychological symptoms in home-dwelling people with dementia: results from the multicomponent cluster randomized controlled LIVE@Home.Path trial. BMC Med. 2022 May 26;20(1):186. doi: 10.1186/s12916-022-02382-5. PMID 35614509
- [Derived] Berge LI, Angeles RC, Gedde MH, Faeo SE, Mannseth J, Vislapuu M, Soyland Puaschitz NG, Hillestad E, Aarsland D, Achterberg WP, Allore H, Ballard C, Li F, Selbaek G, Vahia IV, Husebo BS. Burden and care time for dementia caregivers in the LIVE@Home.Path trial. Alzheimers Dement. 2025 Mar;21(3):e14622. doi: 10.1002/alz.14622. PMID 40042468
- [Derived] Vislapuu M, Patrascu M, Allore H, Husebo BS, Kjerstad E, Gedde MH, Berge LI. Feedback System Analysis of a Multicomponent Intervention on Dyads of Home-Dwelling Persons With Dementia and Their Caregivers: Results From the LIVE@Home.Path Trial. Innov Aging. 2024 Feb 23;8(3):igae020. doi: 10.1093/geroni/igae020. eCollection 2024. PMID 38550899
- [Derived] Puaschitz NGS, Jacobsen FF, Berge LI, Husebo BS. Access to, use of, and experiences with social alarms in home-living people with dementia: results from the LIVE@Home.Path trial. Front Aging Neurosci. 2023 May 22;15:1167616. doi: 10.3389/fnagi.2023.1167616. eCollection 2023. PMID 37284020
- [Derived] Berge LI, Gedde MH, Torrado Vidal JC, Husebo B, Hynninen KM, Knardal SE, Madso KG. The acceptability, adoption, and feasibility of a music application developed using participatory design for home-dwelling persons with dementia and their caregivers. The "Alight" app in the LIVE@Home.Path trial. Front Psychiatry. 2022 Aug 18;13:949393. doi: 10.3389/fpsyt.2022.949393. eCollection 2022. PMID 36061298
- [Derived] Gedde MH, Husebo BS, Vahia IV, Mannseth J, Vislapuu M, Naik M, Berge LI. Impact of COVID-19 restrictions on behavioural and psychological symptoms in home-dwelling people with dementia: a prospective cohort study (PAN.DEM). BMJ Open. 2022 Jan 24;12(1):e050628. doi: 10.1136/bmjopen-2021-050628. PMID 35074810
- See also: Protocol — https://pubmed.ncbi.nlm.nih.gov/32517727/
- See also: Access to and interest in assistive technology for home-dwelling people with dementia during the COVID-19 pandemic (PAN.DEM) — https://pubmed.ncbi.nlm.nih.gov/33416012/
- See also: Which factors increase informal care hours and societal costs among caregivers of people with dementia? A systematic review of Resource Utilization in Dementia (RUD). — https://pubmed.ncbi.nlm.nih.gov/34536149/
- See also: Factors associated with access to assistive technology and telecare in home-dwelling people with dementia: baseline data from the LIVE@Home.Path trial — https://pubmed.ncbi.nlm.nih.gov/34525979/
- See also: The consequences of COVID-19 lockdown for formal and informal resource utilization among home-dwelling people with dementia: results from the prospective PAN.DEM study — https://pubmed.ncbi.nlm.nih.gov/34551783/
- See also: Intensive Medicine and Nursing Home Care in Times of SARS CoV-2: A Norwegian Perspective — https://pubmed.ncbi.nlm.nih.gov/32381282/
- See also: Sensing Technology to Monitor Behavioral and Psychological Symptoms and to Assess Treatment Response in People With Dementia — https://pubmed.ncbi.nlm.nih.gov/32116687/
- See also: The Impact of Deprescribing Psychotropic Drugs on Behavioral and Psychological Symptoms and Daily Functioning in Nursing Home Patients — https://pubmed.ncbi.nlm.nih.gov/32753339/
- See also: Fæø SE, Bruvik FK, Tranvåg O, Husebo BS. Home-dwelling persons with dementia's perception on care support — https://pubmed.ncbi.nlm.nih.gov/31986964/
- See also: The compound role of a coordinator for home-dwelling persons with dementia and their informal caregivers: qualitative study — https://pubmed.ncbi.nlm.nih.gov/33198779/
- See also: We live as good a life as we can, in the situation we're in" - the significance of the home as perceived by persons with dementia. — https://pubmed.ncbi.nlm.nih.gov/31170916/
- See also: The impact of medication reviews by general practitioners on psychotropic drug use and behavioral and psychological symptoms in home-dwelling people with dementia: results from the multicomponent cluster randomized controlled LIVE@Home.Path trial — https://pubmed.ncbi.nlm.nih.gov/35614509/

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT04043364/SAP_000.pdf